CLINICAL TRIAL: NCT02909192
Title: Bright Light Modulation of Non-motor Symptoms in Parkinson's Disease
Brief Title: Bright Light Therapy for Non-motor Symptoms in Parkinson's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Aleksandar Videnovic, MD, Assistant Neurologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016P001775
Record Dates: First submitted 2016-09-15; First posted 2016-09-21 (Estimated); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Excessive Daytime Sleepiness; Circadian Rhythms; Light Therapy
MeSH Terms: conditions — Parkinson Disease; Disorders of Excessive Somnolence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Bright light therapy (Active Comparator): Participants will be treated twice daily with bright light therapy.
  Interventions: Device: Light Therapy Device
- Dim-Red light therapy (Active Comparator): Participants will be treated twice daily with dim-red light therapy.
  Interventions: Device: Light Therapy Device

INTERVENTIONS:
Device: Light Therapy Device

SUMMARY:
Disruption of sleep and alertness is one of the most disabling non-motor symptoms of Parkinson's disease (PD). Mechanisms leading to impaired sleep and alertness in PD are not well understood, and treatment options remain limited. The proposed research will examine markers of the circadian system, sleepiness and sleep quality in PD patients. Further, the project will examine effects of bright light exposure on circadin function, sleep and alertness in PD.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of idiopathic PD as defined by the United Kingdom PD Society Brain Bank Criteria
2. PD Hoehn and Yahr stage 2-4
3. Pittsburgh Sleep Quality Index (PSQI) score ≥ 5
4. Treatment with levodopa and/or dopamine agonist; adjunctive PD medications will be allowed
5. Stable dose of PD medications for at least 4 weeks prior to the study screening.

Exclusion criteria:

1. Atypical or secondary forms of parkinsonism
2. Co-existent significant sleep apnea (as assessed by polysomnography- derived apnea/hypopnea index ≥15 events/hr of sleep)
3. Co-existent restless legs syndrome (RLS), as assessed by the International Classification of Sleep Disorders (ICDS) diagnostic criteria for RLS
4. Cognitive impairment as determined by the Mini-Mental State Examination (MMSE) score of ≤ 26
5. Presence of depression defined as the Beck Depression Inventory (BDI) score >14
6. Untreated hallucinations or psychosis (drug-induced or spontaneous)
7. Use of hypno-sedative drugs for sleep or stimulants; participants will be allowed to taper these drugs and will become eligible 4 weeks after the taper is completed
8. Use of Selective Serotonin Reuptake Inhibitors (SSRIs) / Serotonin-Norepinephrine Reuptake Inhibitors (SNRIs) antidepressants, unless the participant has been on a stable dose for at least 3 months prior to the screening
9. Use of medications known to affect melatonin secretion, such as lithium, alpha- and beta-adrenergic antagonists
10. Shift work, currently or within the prior 3 months
11. Travel through ≥ 2 time zones within 60 days prior to study screening
12. Hematocrit <32 mm3
13. Pre-existing glaucoma/retinal disease contraindicated for light therapy (LT)
14. Dense cataracts
15. Use of medications known to photosensitize retinal tissue (phenothiazines, chloroquine, amiodarone, St. John's Wort)
16. Unstable/serious medical illness.
17. Pregnancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2016-12; Primary Completion 2022-07-05 (Actual); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Parkinson's Disease Sleep Scale (PDSS-2) score to measure sleep quality | 8 weeks

SECONDARY OUTCOMES:
Epworth Sleepiness Scale (ESS) score to measure daytime sleepiness | 8 weeks
Non-Motor Symptoms Assessment Scale for Parkinson's Disease (NMSS) score to measure the severity and frequency of non-motor symptoms | 8 weeks
Plasma melatonin levels collected through blood samples to measure melatonin amplitude and circadian regulation | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandar Videnovic, MD, MSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided